CLINICAL TRIAL: NCT01107223
Title: Long Term Effect of General Practitioner Education on Antibiotic Prescribing: a Large Scale Randomized Study
Brief Title: Long Term Effect of General Practitioner Education on Antibiotic Prescribing
Acronym: PAAIR2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Henri Mondor University Hospital (Other)
Responsible Party: Pr Claude Attali, Henri Mondor University Hospital, department of General Practice
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PAAIR2
Record Dates: First submitted 2010-03-04; First posted 2010-04-20 (Estimated); Last update posted 2010-04-20 (Estimated); Status verified 2010-02

CONDITIONS: Respiratory Tract Infections
Keywords: Antibiotic; Prescribing behaviour; Guidelines; Respiratory tract infections; Non-antibiotic prescription
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Training to antibiotic prescription (Experimental): Physicians randomized in the education group attended a two days seminar focussed on evidence-based guidelines on antibiotic use in respiratory tract infections.
  Interventions: Other: Experimental: Training to antibiotic prescription
- control (Placebo Comparator)
  Interventions: Other: No education on antibiotic prescription rules.

INTERVENTIONS:
Other: Experimental: Training to antibiotic prescription — GPs assigned to the intervention group attended a two days didactic educational meeting on evidence-based guidelines for diagnosis and treatment of acute respiratory tract infection.
  Arms: Training to antibiotic prescription
Other: No education on antibiotic prescription rules. — GPs assigned to control group received no specific recommendations on antibiotic prescription.
  Arms: control

SUMMARY:
Respiratory tract infections are the most common indication for antibiotic prescribing in primary care. Several studies have shown a strong relationship between antibiotic use and bacterial resistance. The aim of this trial was to assess the long-term effect of a continuous education program on general practitioners antibiotic prescribing behaviour. 170 physicians were included in this study. Physicians randomized in the education group attended a two days seminar focused on evidence-based guidelines on antibiotic use in respiratory tract infections. The intervention was limited at physicians level and did not target the patients.

ELIGIBILITY:
Inclusion Criteria:

* General practitioners practicing in three departments of the Parisian area in France
* General practitioners attending a two days didactic educational meeting on evidence-based guidelines for diagnosis and treatment of acute respiratory tract infection.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2004-09; Primary Completion 2009-04 (Actual); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Change in the percentage of prescriptions containing an antibiotic between control and intervention groups (seminar on the treatment of respiratory tract infections). | Effect of the intervention 4 to 6 months after the educational training.
  All prescriptions written by all general practitioners enrolled in the study were extracted each year from the French National Health System database. All data were compared to 2004 (baseline). Education group GPs attended a two-day seminar presenting evidence-based guidelines on antibiotic prescription in respiratory tract infections. The change (compared to baseline) in the percentage of prescriptions containing an antibiotic (antibiotic prescription rates) was compared between control and intervention groups.
Change in the cost of antibiotic prescription between control and intervention groups (seminar on the treatment of respiratory tract infections). | Effect of the intervention 4 to 6 months after the educational training.
  All prescriptions written by all general practitioners enrolled in the study were extracted each year from the French National Health System database. All data were compared to 2004 (baseline). Education group GPs attended a two-day seminar presenting evidence-based guidelines on antibiotic prescription in respiratory tract infections. The change (compared to baseline) in the cost of antibiotic prescription was compared between control and intervention groups.

SECONDARY OUTCOMES:
Long term antibiotic prescription rates | Effect of the intervention 28 to 30 months after the educational training.
  Long term change in the percentage of antibiotic prescriptions between both groups
Long term antibiotic cost. | Effect of the intervention 28 to 30 months after the educational training.
  Long term change in the cost of antibiotic prescriptions between both groups
Symptomatic drug prescription rates | Effect of the intervention 28 to 30 months after the educational training.
  Prescription rates of symptomatic drug for respiratory infections between both groups
Symptomatic drug cost. | Effect of the intervention 28 to 30 months after the educational training.
  Cost of symptomatic drug between both groups
Effect of patient age. | Effect of the intervention 28 to 30 months after the educational training.
  Effect of patient age on antibiotic prescription between both groups
Effect of a seminar on problem-solving strategy on prescriptions. | Effect of the intervention 28 to 30 months after the educational training.
  A second randomization was performed among the intervention group. In one subgroup, GPs attended an additional seminar on problem-solving strategies. Antibiotic prescription rates were compared between controls, evidence-based and problem-solving subgroups. Antibiotic cost was also compared between the both subgroups

CONTACTS AND LOCATIONS:
Overall Officials: Clause Attali, MD, Principal Investigator — Henri Mondor University Hospital
Locations (1):
- Henri Mondor Hospital, department of general practice, Créteil, France

REFERENCES:
- [Derived] Ferrat E, Le Breton J, Guery E, Adeline F, Audureau E, Montagne O, Roudot-Thoraval F, Attali C, Le Corvoisier P, Renard V. Effects 4.5 years after an interactive GP educational seminar on antibiotic therapy for respiratory tract infections: a randomized controlled trial. Fam Pract. 2016 Apr;33(2):192-9. doi: 10.1093/fampra/cmv107. Epub 2016 Jan 21. PMID 26797464